CLINICAL TRIAL: NCT03594552
Title: Modulation of the Brain Excitatory/Inhibitory (E/I) Balance Through Neuronal and Glial Systems in Autism Spectrum Disorder (ASD
Brief Title: Modulation of the Brain Excitatory/Inhibitory (E/I) Balance in Autism Spectrum Disorder (ASD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Principal Investigator, Dr Grainne McAlonan, Deputy head of department, King's College London
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: HR16-17 4081
Record Dates: First submitted 2018-06-27; First posted 2018-07-20 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; Arbaclofen; E-I balance; pharmacological imaging; GABA
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: Repeated-measures cross-over study, where each subject received each one of the three pharmacological probes in separate visits (i.e., placebo, arbaclofen low dose and arbaclofen high dose), with the order of tablet administration being pseudorandomized.
Who Masked: Participant, Investigator
Masking Description: Participants and investigators were blinded to the drug condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Placebo, Arbaclofen_15, Arbaclofen_30 (Experimental): Dose order: Placebo, Arbaclofen 15mg, Arbaclofen 30mg
  Interventions: Drug: Arbaclofen_15; Drug: Arbaclofen_30; Drug: Placebo
- Placebo, Arbaclofen_30, Arbaclofen_15 (Experimental): Dose order: Placebo, Arbaclofen 30mg, Arbaclofen 15 mg
  Interventions: Drug: Arbaclofen_15; Drug: Arbaclofen_30; Drug: Placebo
- Arbaclofen_30, Placebo, Arbaclofen_15 (Experimental): Dose order: Arbaclofen 30mg, Placebo, Arbaclofen 15mg
  Interventions: Drug: Arbaclofen_15; Drug: Arbaclofen_30; Drug: Placebo
- Arbaclofen_15, Placebo, Arbaclofen_30 (Experimental): Dose order: Arbaclofen 15mg, Placebo, Arbaclofen 30mg
  Interventions: Drug: Arbaclofen_15; Drug: Arbaclofen_30; Drug: Placebo
- Arbaclofen_15, Arbaclofen_30, Placebo (Experimental): Dose order: Arbaclofen 15mg, Arbaclofen 30mg, Placebo
  Interventions: Drug: Arbaclofen_15; Drug: Arbaclofen_30; Drug: Placebo
- Arbaclofen_30, Arbaclofen_15, Placebo (Experimental): Dose order: Arbaclofen 30mg, Arbaclofen 15mg, Placebo
  Interventions: Drug: Arbaclofen_15; Drug: Arbaclofen_30; Drug: Placebo

INTERVENTIONS:
Drug: Arbaclofen_15 — Single oral dose (15mg)
  Other Names: r-baclofen, STX209
Drug: Arbaclofen_30 — Single oral dose (30mg)
  Other Names: r-baclofen, STX209
Drug: Placebo — Single oral dose placebo (oral tablet)
  Other Names: Placebo oral tablet

SUMMARY:
This study investigates the brain response to a single acute dose of Arbaclofen, the R-enantiomer of the GABA-B agonist Baclofen, compared to a single dose of placebo in healthy men with and without autism spectrum disorder.

DETAILED DESCRIPTION:
Previous research suggests that GABAergic drug compounds could shift brain excitation and inhibition (E-I) in the healthy brain and in neurodevelopmental psychiatric conditions, such as autism spectrum disorder (ASD) - where this balance is disrupted. A study by Ajram et al. (2017) has shown an E-I shifted towards more GABA in individuals with ASD, and not in controls, after a single dose of the anti-glutamatergic and pro-GABAergic drug Riluzole. Moreover, brain connectivity patterns in ASD patients where shifted towards the ones observed in the control group. However, it was unclear whether this changes could be driven by GABA receptors, thus more specific probes may help to clarify the mechanism underlying the E-I coordination in ASD. Therefore, this study will use neuroimaging and electrophysiology to investigate the brain E-I coordination in ASD compared to control participants when the system is responding to a single dose of the specific GABA-B (STX209) receptor agonist. 50 adult individuals with ASD and 50 neurotypical adults (25 males and 25 females per group) will be invited to participate. Each participant will receive a single dose of the drug (15mg or 30mg Arbaclofen) or matched placebo). Brain activity and neurochemistry will be investigated using magnetic resonance imaging. Further data will be collected through questionnaires, behavioural tasks, blood samples, and sensory tasks using electroencephalography and retinal imaging.

ELIGIBILITY:
Inclusion Criteria:

* ASD participants must pass diagnostic threshold for ASD on the Autism Diagnostic Interview-Revised (if and informant is available)
* ASD participants must be currently symptomatic on Autism Diagnostic Observation Schedule (ADOS)
* Age 18-60 years
* Can give informed consent
* medication free in the month preceding participation; but regular medication (used in a stable dose over the two months previous to participation) with drug which does not affect glutamate or GABA directly may be permitted
* IQ>70

Exclusion Criteria:

* IQ<70
* history of psychosis, co-morbid major mental illness, significant physical illness (heart disease, high blood pressure, seizures) habitual substance misuse (including alcohol)
* ASD caused by a known genetic syndrome e.g. Fragile X or 22q11 deletion syndrome,
* past/present treatment for epilepsy
* Change of medication dose/start of a new pharmacological therapy in the month prior to participation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Neurochemical response to GABAergic stimulation. | Through study completion, an average of 2 years.
  Comparing brain excitation-inhibition measures (i.e., glutamate and GABA) when the GABAergic system is activated by a single oral dose of the GABA-B drug Arbaclofen versus the placebo condition.

SECONDARY OUTCOMES:
Functional connectivity measures using resting state functional magnetic resonance imaging. | Through study completion, an average of 2 years.
  Maps of functional connectivity will be obtained for each condition and compared between adults with and without ASD.
Brain oscillations under sensory stimulation | Through study completion, an average of 2 years.
  Brain oscillations and event-related potentials will be recorded during sensory stimulation using high density electroencephalography.

CONTACTS AND LOCATIONS:
Overall Officials: Grainne McAlonan, PhD, Principal Investigator — King's College London
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No